CLINICAL TRIAL: NCT01594723
Title: A Phase 2 Study of LY2784544 in Patients With Myeloproliferative Neoplasms
Brief Title: A Study of LY2784544 in Participants With Myeloproliferative Neoplasms
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13861; I3X-MC-JHTB (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-05-01; First posted 2012-05-09 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Neoplasms, Hematologic
MeSH Terms: conditions — Hematologic Neoplasms | interventions — LY2784544

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 120 mg LY2784544 (Experimental): 120 milligram (mg) administered orally once daily for 6 cycles (168 days)
  Interventions: Drug: 120 mg LY2784544

INTERVENTIONS:
Drug: 120 mg LY2784544 — Administered orally

SUMMARY:
The primary purpose of this study is to measure the response rate in participants with the myeloproliferative neoplasms (MPNs), polycythemia vera (PV), essential thrombocythemia (ET), or myelofibrosis (MF) when treated with LY2784544, including those who have demonstrated an intolerance to, failure of primary response to, or have demonstrated disease progression while on ruxolitinib.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of polycythemia vera (PV), essential thrombocythemia (ET), or myelofibrosis (MF) as defined by the World Health Organization (WHO) diagnostic criteria for myeloproliferative neoplasms (Swerdlow et al. 2008) and meet the following additional subtype specific criteria:

  * PV: have failed or is intolerant of standard therapies or refuses to take standard medications
  * ET: have failed or is intolerant of standard therapies or refuses to take standard medications
  * MF (participants with MF must meet at least 1 of the following): have intermediate 1, intermediate 2, or high-risk MF according to the Dynamic International Prognostic Scoring System (DIPPS Plus) for Primary Myelofibrosis (Gangat et al. 2011); or have symptomatic MF with spleen greater than 10 centimeter (cm) below left costal margin; or have post-polycythemic MF; or have post-ET MF
* All PV, ET, and MF participants must meet the following criteria:

  o Have a quantifiable level of janus kinase 2 with a valine to phenylalanine substitution at amino acid 617 (JAK2 V617F) mutation. This inclusion criterion will not apply to the subset of participants in Cohorts 10 and 11 that must be negative for the JAK2 V617F mutation
* Are ≥ 18 years of age
* Have given written informed consent prior to any study-specific procedures
* Have adequate organ function, including: Hepatic: Direct bilirubin ≤1.5 times upper limits of normal (ULN), alanine transaminase (ALT), and aspartate transaminase (AST) ≤2.5 times ULN; Renal: Serum creatinine ≤1.5 times ULN; Bone Marrow Reserve: Absolute neutrophil count (ANC) ≥1000/microliter (mcL), platelets ≥50,000/mcL for participants with ET or PV and ≥25,000/mcL for participants with MF
* Have a performance status of 0, 1, or 2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued all previous approved therapies for Myeloproliferative Neoplasms (MPNs), including any chemotherapy, immunomodulating therapy (for example, thalidomide, interferon-alpha), immunosuppressive therapy (for example, corticosteroids >10 mg/day prednisone or equivalent), radiotherapy, and erythropoietin, thrombopoietin, or granulocyte colony stimulating factor for at least 14 days and recovered from the acute effects of therapy. Hydroxyurea used to control blood cell counts is permitted at study entry if the subject has been maintained on a stable dose for at least 4 weeks. Low-dose acetylsalicylic acid (aspirin) is permitted as well
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the study and for 3 months following the last dose of study drug
* Females with child-bearing potential must have had a negative urine pregnancy test ≤ 7 days before the first dose of study drug and must also not be breastfeeding
* Are able to swallow capsules
* For participants who have undergone recent major surgery, at least 28 days must have elapsed between surgery and study participation and the participant must have achieved, in the opinion of the treating physician, at least a good recovery from the surgical procedure
* Enrollment into Cohort 12 is limited to MF, PV, or ET participants, regardless of mutational status, who, in addition to all other criteria, have demonstrated intolerance to ruxolitinib, failure of primary response to ruxolitinib, or have demonstrated disease progression while on ruxolitinib

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 14 days from a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have a corrected QT (QTc) interval >470 millisecond (msec) using Bazett's formula
* Have serious preexisting medical conditions that, in the opinion of the investigator would preclude participation in the study (for example a gastrointestinal disorder causing clinically significant symptoms such as nausea, vomiting, and diarrhea, or malabsorption syndrome)
* Are currently being treated with agents that are metabolized by Cytochrome P450 3A4 enzyme (CYP3A4) with a narrow therapeutic margin (for example, alfentanil, cyclosporine, diergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, and tacrolimus) or Cytochrome P450 2B6 enzyme (CYP2B6) (for example, cyclophosphamide, ifosfamide, tamoxifen, efavirenz, propofol, methadone, and bupropion)
* Are currently being treated with warfarin or one of its derivatives which is known to alter levels of protein C or protein S. An exception to this criterion will be allowed for participants with a prior history of Budd-Chiari Syndrome who are being treated with warfarin or one of its derivatives
* Have received a hematopoietic stem cell transplant
* Have a second primary malignancy that in the judgment of the Investigator and Sponsor may affect the interpretation of results
* Have an active fungal, bacterial, and/or known viral infection including human immunodeficiency virus (HIV) or viral (A, B, or C) hepatitis (screening is not required)
* Have a history of congestive heart failure with New York Heart Association (NYHA) Class >2 (NYHA Class 1 and 2 are eligible), unstable angina, recent myocardial infarction (within 6 months prior to administration of study drug), or documented history of ventricular arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2012-05-22 (Actual); Primary Completion 2015-03-20 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with an Objective Response (Objective Response Rate) | Baseline until Disease Progression (PD) or Participant Stops Study (Estimated up to 24 Months)

SECONDARY OUTCOMES:
Percentage of Participants with a Molecular Response (Molecular Response Rate) | Baseline until PD or Participant Stops Study (Estimated up to 24 Months)
Percentage of Participants with Hematological Improvement (Hematological Improvement Rate) | Baseline until PD or Participant Stops Study (Estimated up to 24 Months)
Change in Spleen Size | Baseline until PD or Participant Stops Study (Estimated up to 24 Months)
Change in Bone Marrow Fibrosis Grade | Baseline until PD or Participant Stops Study (Estimated up to 24 Months)
Change in Number of Thrombotic or Hemorrhagic Events | 3 Months prior to Study Drug (historic) until PD or Participant Stops Study (Estimated up to 24 Months)
Change in Number of Phlebotomies and Transfusions | Baseline until PD or Participant Stops Study (Estimated up to 24 Months)
Duration of Response | Confirmed Response to PD or Death from Any Cause (Estimated up to 24 Months)
Time to Best Response | Baseline to Confirmed Response (Estimated up to 6 Months)
Change in Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) | Baseline until PD or Participant Stops Study (Estimated up to 24 Months)
Time to Treatment Failure | Baseline to PD, Death from Any Cause or Participant Stops Study (Estimated up to 24 Months)
Time to Disease Progression | Baseline to Measured PD (Estimated up to 24 Months)
Progression Free Survival (PFS) | Baseline to PD or Death from Any Cause (Estimated up to 24 Months)
Change in Activities of Daily Living (ADL)/ Instrumental Activities of Daily Living (IADL) | Baseline until PD or Participant Stops Study (Estimated up to 24 Months)
Change in EuroQol - 5 dimensions (EQ-5D) Index Score | Baseline until PD or Participant Stops Study (Estimated up to 24 Months)
Change in International Prognosis Scoring System Scales (IPSS) | Baseline until PD or Participant Stops Study (Estimated up to 24 Months)
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY2784544 | Predose up to Day 84
PK: Time of Maximal Concentration (Tmax) of LY2784544 | Predose up to Day 84
Change in Liver Size | Baseline until PD or Participant Stops Study (Estimated up to 24 Months)
Change in 6-item Physician Symptom Assessment | Baseline until PD or Participant Stops Study (Estimated up to 24 Months)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLilly (1-877-285-4559) or 1-317-615-4559 Mon- Fri 9 AM - 5 PM Eastern time (UTC/GMT -5 hours, EST), Study Director — Eli Lilly and Company
Locations (39):
- United States (23):
  - Highlands Oncology Group - Duplicate 2, Rogers, Arkansas
  - Providence St. Joseph's Medical Center, Burbank, California
  - Norwalk Hospital, Norwalk, Connecticut
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Palm Beach Cancer Institue, West Palm Beach, Florida
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Indiana Blood & Marrow Transplantation (IBMT), Indianapolis, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University Medical Center, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Weill Cornell Medical College, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Mid Ohio Oncology Hematology, Columbus, Ohio
  - Baptist Cancer Center, Memphis, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Joe Arrington Cancer Center, Lubbock, Texas
  - Swedish Medical Center, Seattle, Washington
  - Dean Medical Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garran, Australian Capital Territory
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wodonga, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perth, Western Australia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Austria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec, Canada
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris, France
- Germany (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minden
- Italy (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
- Sweden (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uddevalla
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uppsala